CLINICAL TRIAL: NCT00978497
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Ascending Multiple Dose Trial of the Safety, Efficacy, and Pharmacokinetics of ANA598 Administered With Pegylated Interferon and Ribavirin in Treatment-Naïve Genotype 1 Patients With Chronic Hepatitis C Infection
Brief Title: Safety, Tolerability, and Antiviral Activity of ANA598 Administered in Combination With Pegylated Interferon and Ribavirin for the Treatment of Genotype-1 Chronic HCV Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ANA598-504
Record Dates: First submitted 2009-09-16; First posted 2009-09-17 (Estimated); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: HCV Infection
MeSH Terms: conditions — Hepatitis C | interventions — setrobuvir; Ribavirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Placebo Comparator): Peginterferon and ribavirin + placebo BID for 12 weeks, followed by Peg-IFN and RBV for an additional 12 or 36 weeks
  Interventions: Drug: placebo; Drug: Peginterferon; Drug: Ribavirin
- 2 (Experimental): ANA598 200 mg BID + Peginterferon and ribavirin for 12 weeks, followed by Peg-IFN and RBV for an additional 12 or 36 weeks
  Interventions: Drug: ANA598; Drug: Peginterferon; Drug: Ribavirin
- 3 (Experimental): ANA598 400mg BID + Peginterferon and ribavirin for 12 weeks, followed by Peg-IFN and RBV for an additional 12 or 36 weeks
  Interventions: Drug: ANA598; Drug: Peginterferon; Drug: Ribavirin

INTERVENTIONS:
Drug: placebo — oral BID
  Arms: 1
Drug: ANA598 — oral 200mg BID
  Arms: 2
Drug: ANA598 — oral 400mg BID
  Arms: 3
Drug: Peginterferon — 180 μg dose via subcutaneous injection weekly
Drug: Ribavirin — oral 1000 mg/day for patients who weighed < 75 kg and 1200 mg/day for patients who weighed ≥ 75 kg

SUMMARY:
The purpose of this study is to assess the safety, tolerability and effectiveness of ANA598 when administered with pegylated interferon and ribavirin (Standard of Care [SOC]) compared to placebo + SOC.

DETAILED DESCRIPTION:
The safety, tolerability and antiviral activity of ANA598, administered orally at 200 mg BID or 400 mg BID for 12 weeks in combination with pegylated interferon and ribavirin (SOC) will be compared to placebo + SOC. Treatment-naïve patients with genotype 1 infection will be eligible for enrollment. Patients randomized to ANA598 will receive a loading dose of 800 mg q 12 hours administered on the first day of dosing. Patients with undetectable HCV RNA at week 4 and week 12 will be randomized to receive either an additional 12 or 36 weeks of SOC alone.

Ninety patients will be randomized into 2 cohorts. The forty-five patients in each cohort will be randomized as 30 active: 15 placebo.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, ages 18 to 65 years
* Documented chronic HCV infection, genotype 1a or 1b
* Treatment-naïve

Exclusion Criteria:

* Female patients who are pregnant or breast-feeding
* Infection with non-genotype 1 HCV
* Previous treatment for HCV infection
* HIV or HBV positive
* Any medical contraindication to Peg-IFN or RBV therapy
* History of any other known cause of liver disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2009-09; Primary Completion 2010-04 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Undetectable HCV RNA | 12 Weeks

SECONDARY OUTCOMES:
Safety and Tolerability | Throughout study
Undetectable HCV RNA | Week 4, Week 24, and Week 48
ANA598, Peg-IFN-a-2-a, ribavirin concentrations | Various time points through Week 12
Undetectable HCV RNA | 24 weeks after completion of therapy for sustained virologic response [SVR]

CONTACTS AND LOCATIONS:
Locations (21):
- United States (20):
  - United States, California 1, Anaheim, California
  - United States, California 4, Los Angeles, California
  - United States, California 2, San Clemente, California
  - United States, California 3, San Diego, California
  - United States, California 5, San Francisco, California
  - United States, Florida 2, Gainesville, Florida
  - United States, Florida 3, Miami, Florida
  - United States, Florida 1, Sarasota, Florida
  - United States, Maryland, Lutherville, Maryland
  - United States, Massachusetts, Boston, Massachusetts
  - United States, Michigan, Detroit, Michigan
  - United States, New York, New York, New York
  - United States, North Carolina, Chapel Hill, North Carolina
  - United States, North Carolina, Durham, North Carolina
  - United States, Ohio, Cincinnati, Ohio
  - United States, Pennsylvania, Philadelphia, Pennsylvania
  - United States, Texas 2, Houston, Texas
  - United States, Texas 1, San Antonio, Texas
  - United States, Virginia 1, Fairfax, Virginia
  - United States, Virginia 2, Falls Church, Virginia
- Puerto Rico, Santurce, Puerto Rico